CLINICAL TRIAL: NCT06739655
Title: Preoperative Radiation Therapy and Immediate Breast Reconstruction, a Phase 3 Randomized Controlled Trial in the Belgian Population
Brief Title: Preoperative Radiation Therapy and Immediate Breast Reconstruction
Acronym: PRADAIIBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Research Antwerp (Other)
Collaborators: Ziekenhuis aan de Stroom (Other); Iridium netwerk (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO23023GZA
Record Dates: First submitted 2024-12-02; First posted 2024-12-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Breast Neoplasms; Breast Carcinoma; Breast Adenocarcinoma; Cancer; Neoplasm
Keywords: Breast cancer; Radiotherapy; PRADA; Breast reconstruction; BreastQ; QoL; Skin Sparing Mastectomy; Mastectomy; Breast surgery; radiation therapy; Preoperative radiation therapy; Preoperative RT; Cosmesis; Breast satisfaction; Immediate Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Multicenter phase 3 (non-pharmacological) randomized controlled trial, with a parallel design and a 1:1 assignment ratio.
Masking Description: This is an open-label study due to the impracticalities and ethical considerations regarding blinding of both radiation therapy and (sham-)surgeries.
  The assessment of the photographs by an external expert panel will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment arm (SoC; PostOperative RT) (Active Comparator): Treatment in this arm consists of:
  1. Mastectomy
  2. Immediate or delayed breast reconstruction.
  3. Postoperative radiation therapy, according to the SoC as indicated by international guidelines.
  [Systemic treatments are not considered as study treatments and will be implemented at the discretion of the treating physician.]
  Interventions: Radiation: Postoperative radiotherapy; Procedure: Immediate or delayed breast reconstruction
- Experimental treatment arm (PreOperative RT) (Experimental): Treatment in this arm consists of:
  1. Preoperative radiation therapy (Preop-RT). Preop-RT will be administered according to the same parameters and quality standards as PMRT/WBRT, as indicated by international guidelines.
  2. Mastectomy combined with immediate breast reconstruction, after a 2-6 weeks interval.
  [Systemic treatments are not considered as study treatments and will be implemented at the discretion of the treating physician.]
  Interventions: Radiation: Preoperative radiotherapy; Procedure: Immediate breast reconstruction

INTERVENTIONS:
Radiation: Preoperative radiotherapy — In this study patients assigned to the experimental treatment arm will receive preoperative radiation therapy instead of postoperative radiation therapy (PMRT).
  This preoperative radiation therapy will be administered according to the standard of care (SoC) principles for PMRT and Whole Breast Radiation Therapy (WBRT) as defined by international guidelines.
  Other Names: Preop-RT; Neoadjuvant radiation therapy; NART
  Arms: Experimental treatment arm (PreOperative RT)
Radiation: Postoperative radiotherapy — Standard of care (SoC) postoperative radiotherapy, as defined by international guidelines.
  Other Names: Postop-RT; Postmastectomy Radiation Therapy; PMRT; Adjuvant Radiation Therapy; ART
  Arms: Standard treatment arm (SoC; PostOperative RT)
Procedure: Immediate breast reconstruction — In the experimental arm of the PRADAIIBE, the participants will undergo immediate breast reconstruction surgery. This is defined as breast reconstruction taking place at the same time as oncological surgery. Using one of the following primary techniques: 1) Autologous tissue reconstruction ; 2) Breast implant based reconstruction; 3) Combined autologous tissue and breast implant reconstruction. These techniques can take place in a single phase, or in a two-phased (tissue expander) approach.
  Adjuvant techniques (e.g.: lipofilling, mesh, ADM etc.) could be added.
  Other Names: IBR
  Arms: Experimental treatment arm (PreOperative RT)
Procedure: Immediate or delayed breast reconstruction — In the standard arm of the PRADAIIBE, the participants will undergo immediate or delayed breast reconstruction surgery. This is defined as breast reconstruction taking place at the same time as oncological surgery (immediate), or at a later time (delayed). Using one of the following primary techniques: 1) Autologous tissue reconstruction ; 2) Breast implant based reconstruction; 3) Combined autologous tissue and breast implant reconstruction. These techniques can take place in a single phase, or in a two-phased (tissue expander) approach. Adjuvant techniques (e.g.: lipofilling, mesh, ADM etc.) could be added.
  Arms: Standard treatment arm (SoC; PostOperative RT)

SUMMARY:
The goal of this phase III randomized controlled trial (PRADAIIBE) is to assess if preoperative radiation therapy (Preop-RT) combined with immediate breast reconstruction (IBR) can safely improve both aesthetic and quality of life outcomes in breast cancer patients, compared to the standard of care (SoC) therapy consisting of post-mastectomy radiation therapy (PMRT) and delayed/immediate breast reconstruction, in a population of breast cancer patients with an indication of mastectomy and PMRT.

The following hypotheses and outcomes will be assessed at the primary endpoint of 1 year of follow-up:

* Efficacy: Does Preop-RT+IBR lead to a higher BREAST-Q satisfaction with breasts score (primary endpoint), EQ-5D-5L VAS score , EQ-5D-5L Index score, AIS-Total Aesthetic Score, or a shorter treatment duration compared to SoC?
* Safety: Does Preop-RT+IBR lead to an increase in adverse events (general or surgical), a lower rate of pathologic Complete Response (pCR), or worse survival outcomes compared to SoC? [Note: this study was not powered as a non-inferiority trial, all outcomes will be pooled internationally with parallel studies]

Eligible and consenting participants will undergo screening and baseline assessments. They will then be randomised between experimental (Preop-RT+IBR) and control (SoC) groups, in a 1:1 stratified variable block size design. Follow-up will take place at 3 months, 1, 2, 5, and 10 years after the last study treatment. At baseline and during each follow-up visit each participant will complete the Breast Q 'satisfaction with breasts' and EQ-5D-5L scales, photographs will be taken. During follow-up pCR will be assessed if applicable, adverse events will be registered, and oncological follow-up will be recorded.

DETAILED DESCRIPTION:
The PRADAIIBE study is a multicentric phase III randomized controlled trial, investigating the effects of radiation therapy timing on breast reconstruction results in breast cancer patients.

This study will recruit adult female breast cancer patients from the Belgian population, who have an indication for mastectomy, Post-Mastectomy Radiation Therapy (PMRT), and also have a wish for breast reconstruction.

After informed consent is signed, patients will be screened, and included in the study if all eligibility criteria are met. If they are not eligible for participation or choose to withdraw after the ICF was signed, they will be registered as a 'screen failure'.

After study inclusion, baseline assessments take place, this includes two questionnaires, one focussed on patient's satisfaction with their own breasts (BREAST-Q v2, BQ-score), the other one focussed on their quality of life perception (EQ-5D-5L VAS-score and Index-score). Next, four photographs of the exposed breast area will be taken. These photographs will later be assessed by an expert panel (AIS-TAS).

Eligible participants are randomized using the central eCRF randomization tool (Castor EDC). Randomisation is stratified on study site and a variable block size will be used. Resulting in random assignment to one of the following treatment arms:

* Control (SoC) treatment arm: Mastectomy followed by PMRT and delayed (or immediate) breast reconstruction.
* Experimental treatment arm: preoperative radiation therapy (preop-RT) followed by mastectomy and immediate breast reconstruction.

Those assigned to the control group will follow the standard of care (SoC) treatment consisting of oncological surgery (within 6 weeks of randomisation or end of preop chemotherapy) followed by radiation therapy (PMRT) within 6-12 weeks. The breast reconstruction surgery will take place either at the same time (e.g. tissue expander implantation) as the oncological surgery, or at a delayed moment (usually a 6-12 months delay).

Patients assigned to the intervention group will receive preop-RT (within 6 weeks of randomisation or end of preop chemotherapy), and after an interval of 2-6 weeks mastectomy combined with immediate breast reconstruction will be performed. The radiation therapy will be administered according to the same principles as PMRT/Whole Breast Radiation Therapy (WBRT). This change to preoperative timing of the radiation therapy allows for immediate breast reconstruction without irradiation of the reconstructed breast.

In the unexpected event of tumour downstaging due to preoperative treatment, changing the indication from mastectomy to breast conserving surgery (BCS), while the patient has already been included, it is allowed within the study protocol to perform BCS. In this case the patient should receive the treatment and surgery which is in their best interest. The same follow-up will be provided. In statistical analysis results from such patients will be handled according to the inter-current events (ICE) strategies defined in the SAP. However, such downstaging is not expected from preop-RT at such a short treatment interval of 2-6 weeks.

Systemic therapy will be administered per standard of care, according to the discretion of the treating medical oncologist. Systemic therapy details will be registered in the eCRF, but it is not considered as part of the study treatments, and will not be manipulated within this trial.

After the treatment period is finished (last study treatment) follow-up will take place at 3 months, 1 year, 2 years, 5 years and 10 years. In the control group, patients undergoing delayed breast reconstruction will be invited to an intermediate follow up visit (IMFU) visit at 3 months after conclusion of radiation therapy. The reason for this IMFU visit is to capture the outcomes of interest in the interval between mastectomy and breast reconstruction, as well as provide continued study follow-up during this long treatment interval of +/- 6-12 months.

During each follow-up visit the BREAST-Q and EQ-5D-5L questionnaires will be assessed, photographs will be taken and evaluated at a later (expert panel using the AIS-tool), adverse events will be elicited, pathologic response assessed, treatment milestones are recorded (treatment duration) and oncological recurrence is assessed from the +1 year visit onwards according to the events and outcomes described in the DATECAN 2015 initiative.

ELIGIBILITY:
Screening assessments, including review of all study eligibility criteria must be completed before enrolment and randomisation.

Inclusion criteria:

In order to be eligible to participate in this study, a participant must meet all of the following criteria:

1. Women ≥18 years with histopathologically confirmed breast cancer who:

1.a. require SSM/NSM for any reason (e.g. extensive disease)

1.b. require postoperative radiation therapy of at least the chest wall

1. c. have a wish for a breast reconstruction
2. An Eastern Cooperative Oncology Group (ECOG) performance status grade ≤ 2
3. Participant is able and willing to provide written informed consent, which includes compliance with and ability to undergo all study procedures, and attend the scheduled follow-up visit(s) per protocol.

Exclusion criteria:

A potential participant who meets any of the following criteria will be excluded from participation in this study:

1. A previous history of breast cancer or irradiation of the chest wall for any other indication, on the other side (ipsilateral). A bilateral SSM/NSM + reconstruction (e.g. in case of a contralateral prophylactic SSM/NSM), or previous contralateral breast cancer disease/treatment, do not fall under this criterium and are thus allowed.
2. Collagen synthesis disease
3. Ongoing pregnancy
4. Actively breastfeeding
5. Smoking at time of inclusion (a history of smoking is allowed but needs to be registered in the eCRF). No interval between smoking cessation and study inclusion is defined, but the reconstructive surgeon needs to be willing to operate the patient using autologous tissue transfer. This generally translates to a smoking cessation of >3months preoperatively.
6. BMI > 35 kg/m2
7. cT4d tumour, metastatic disease or any reason making SSM/NSM not indicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2029-02-20 (Estimated); Study Completion 2038-02-20 (Estimated)

PRIMARY OUTCOMES:
Patient's satisfaction with breasts. | Measured at 3 months, 1year, 2 years, 5 years and 10 years after last locoregional treatment. Primary endpoint: 1 year after LST.
  Operationalisation (measurement variable):
  The satisfaction with breasts outcome variable is operationalised through the "satisfaction with breasts" scale from the BREAST-Q (v2) 'Reconstruction', 'Breast Conserving Treatment', or 'Mastectomy' modules (as applicable). The answers from the questionnaire are then transformed into a 'BREAST-Q Score', using the provided conversion scales.(3) The BREAST-Q score can range from 0 to100.
  Analysis metric:
  The transformed value of the BREAST-Q score will be used for analysis.
  Method of aggregation:
  Mean, SD, median, IQR, and range will be reported. For comparisons and estimands, please refer to the SAP.

SECONDARY OUTCOMES:
Quality of Life (EQ-5D-5L VAS score) | A baseline assessment is performed during the screening visit, followed by repeated measurements during the IMFU (if applicable), 3M, 1Y, 2Y, 5Y, and 10Y follow-up visits.
  Operationalisation (measurement variable):
  'Quality of Life' will be assessed using the EQ-5D-5L questionnaire. Deriving the VAS-score from the VAS-scale Range EQ-5D-5L VAS-score: 0-100
  Analysis metric:
  The VAS-score will be used as recorded.
  Method of aggregation:
  Mean, SD, median, IQR, and range will be reported. For comparisons and estimands, please refer
Quality of Life (Index score) | A baseline assessment is performed during the screening visit, followed by repeated measurements during the IMFU (if applicable), 3M, 1Y, 2Y, 5Y, and 10Y follow-up visits.
  Operationalisation (measurement variable):
  'Quality of Life' will be assessed using the EQ-5D-5L questionnaire. The index score is calculated from the Likert-scale answers, using a formula validated in the Belgian population.
  Range EQ-5D-5L Index-score: -0.533-0.962.
  Analysis metric:
  The Index-score will be transformed to a scale between 0 and 1, proportional to its original distribution using the following formula:
  F(IS) = (IS+0.533)/1.495 The rationale for this transformation, is to adhere to the scale proposed by the EQ-5D-5L documentation, and improve interpretability.
  Method of aggregation:
  Mean, SD, median, IQR, and range will be reported. For comparisons and estimands, please refer
Breast cosmesis, objective assessment (AIS - TAS) | Photographs are taken during the screening visit, followed by repeated photographs during the IMFU (if applicable), 3M, 1Y, 2Y, 5Y, and 10Y follow-up visits. Expert panel assessment will take place at a later moment.
  Operationalisation (measurement variable):
  Breast cosmesis will be assessed through a blinded panel of experts, using the 'Aesthetic Items Scale' to score a set of photographs taken during study visits. This set will consist of 4 2D digital photographs. The AIS has 5 items, each are scored from 1 to 5. These items are then summed to derive the 'Total Aesthetic Score' (TAS). The TAS can range from 5 to 25.
  Analysis metric:
  The derived value of the Total Aesthetic Score (TAS) from each assessor will be averaged to derive the TAS of each set of photos.
  Method of aggregation:
  Mean, SD, median, IQR, and range will be reported. For comparisons and estimands, please refer to the SAP.
Frequency and severity of adverse events (General AEs) | AEs will be assessed and recorded continuously, with explicit querying during all follow-up visits.
  During the study all adverse events (AEs) codes and grades will be recorded in the eCRF, based on the 'National Cancer Institute Common Terminology Criteria for Adverse Events' (NCI-CTCAE) v5.0 reporting system.
  Analysis metric:
  Tabulation of AE frequency, type and severity. As well as the highest grade AE for each participant.
  Method of aggregation:
  AEs will be aggregated based on their grades. Two composite measures will be reported, consisting of 1) any AE vs. no AE, and 2) grade > 3 AEs vs. no or grade <3 AEs. Tables presenting both frequency and proportions of each grade and the composite measures will be presented. Proportions will be reported as AEs compared to 'highest grade per patient', and to 'total set of AEs'. For comparisons and estimands, please refer to the SAP.
Frequency and severity of adverse events (Surgical AEs) | AEs will be assessed and recorded continuously, with explicit querying during all follow-up visits.
  During the study all adverse events (AEs) codes and grades will be recorded in the eCRF, based on the 'National Cancer Institute Common Terminology Criteria for Adverse Events' (NCI-CTCAE) v5.0 reporting system. ). The relationship to surgical study interventions will be registered in the eCRF.
  Analysis metric:
  Tabulation of surgical AE frequency, type and severity. As well as the highest grade surgical AE for each participant.
  Method of aggregation:
  Surgical AEs will be aggregated based on their grades. Two composite measures will be reported, consisting of 1) any AE vs. no AE, and 2) grade > 3 AEs vs. no or grade <3 AEs, relating to surgical AEs. Tables presenting both frequency and proportions of each grade and composite measures will be presented. Proportions will be reported as surgical AEs compared to 'highest grade per patient', and to 'total set of surgical AEs'. For comparisons and estimands, please refer to the SAP.
Treatment duration | These outcome variables will be continuously recorded as the participant progresses through the study and the data is entered in the eCRF.
  Operationalisation (measurement variable):
  The dates of diagnostic, study, and treatment milestones will be recorded in the eCRF. Time intervals expressed in days, will be assessed for:
  * Randomisation to last study treatment (LST)
  * Randomisation to oncological breast surgery
  * Oncological breast surgery to last study treatment (LST)
  Analysis metric:
  The 'randomisation to last study treatment (LST)' time interval, expressed in days.
  Method of aggregation:
  KM-estimates and derived estimates for central tendency and spread will be provided. For comparisons and estimands, please refer to the SAP
Pathological complete response rate (pCR) | This outcome variable will be assessed after the pathology report of the removed breast tissues is available. This is checked intermittently during the treatment phase, or at least during the 3 months follow-up visit.
  Operationalisation (measurement variable):
  Patients receiving preoperative therapy undergo pathological response assessment of the removed breast tissues (SoC assessment). The reported response Pinder-classification or 'No preoperative therapy' will be recorded in the eCRF.
  Analysis metric:
  The response category as described in the pathology report will be recorded for all participants, but this outcome will only be assessed in participants receiving preoperative-systemic therapy (with, or without Preop-RT).
  This is due to the fact that no response is expected at 2-6 weeks after radiation therapy monotherapy, which would result in an unfair comparison.
  Both this subset of the ITT set, and the complete safety set will be used in the safety assessment, as described in the SAP.
  Method of aggregation:
  The frequency and proportion of the response categories will be presented in a table. For comparisons and estimands, please refer to the SAP.

OTHER OUTCOMES:
Oncological survival and time-to-event data | Oncological TTE data will be registered at 1, 2, 5, and 10 years of follow-up after the last study treatment (LST). However, the exact dates of diagnosis/death will be used.
  Operationalisation (measurement variable):
  The oncological survival and TTE data are operationalised as time-to-event intervals for the events of interest listed below. These events are recorded according to the 2015 DATECAN consensus.
  The following TTE/survival metrics will be reported according to the 2015 DATECAN consensus: Overall Survival (OS), Breast Cancer-Specific Survival (BCSS), Relapse-Free Survival (RFS), Locoregional Relapse-Free Survival (L-RFS), and Distant-Relapse Free Survival (D-RFS).
  Analysis metric:
  The TTE data is registered in days from randomisation (Rz). Censoring will be used for participants without events at the end of their follow up.
  Method of aggregation:
  KM-estimates with derived estimates for central tendency and spread, as well as proportions free from events at follow-up visit timepoints will be reported. The non-aggregated data will be used for survival analysis. For comparisons and estimands, please refer to the SAP.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Machiels, MD, PhD, Principal Investigator — Iridium netwerk
Locations (6):
- Belgium (6):
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem, Antwerpen
  - Ziekenhuis aan de stroom, Wilrijk, Antwerpen
  - AZ Klina, Brasschaat, Antwerp
  - CHU Namur, Namur, Namur
  - Universitair Ziekenhuis Gent (UZGent), Ghent, Oost Vlaanderen
  - AZ Groeninge, Kortrijk, West Vlaanderen

IPD SHARING:
Plan to Share IPD: Yes
All data generated during this study will be anonymised and then shared with the UK based PRADA-consortium and the Dutch BRENAR study (parallel pilot study).
  This PRADA-consortium oversees the organisation of similar trials in other countries, with the goal of publishing the results from these international studies as pooled data in order to increase the sample size and thereby the statistical power of the conclusions.
  Special care will be taken to anonymise all personal data and to adhere with both Belgian and European data protection and privacy laws (GDPR).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared after assessment of the primary endpoint, and subsequently at an interval in accordance with the further follow-up visits.
Access Criteria: Access to the finalised database can be requested after primary endpoint assessment. Requests will be handled on a case-by-case basis. Data will only be shared for scientific purposes, and is only permitted after ethical commission approval, and DTA signing.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT06739655/Prot_SAP_002.pdf